CLINICAL TRIAL: NCT05212129
Title: Hypermobile Ehlers-Danlos Syndrome: Efficacy of Non-invasive Vagal Nerve Stimulation and Effects on Brain-Gut Physiology
Brief Title: Auricular Vagal Nerve Stimulation for Hypermobile Ehlers-Danlos Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University College, London (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Katja Karrento, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1541191
Record Dates: First submitted 2021-11-02; First posted 2022-01-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Functional Gastrointestinal Disorders; Hypermobile Ehlers-Danlos Syndrome; Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Disease; Autonomic Nervous System Imbalance
MeSH Terms: conditions — Gastrointestinal Diseases; Ehlers-Danlos syndrome type 3; Postural Orthostatic Tachycardia Syndrome | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants enrolled in either Treatment Arm A (randomized to active vs sham therapy) or Treatment Arm B at the same time throughout the enrollment process.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment Arm A is masked (double-blinded). Treatment Arm B is not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Arm A (hEDS) (Active Comparator): (n=60) patients who meet criteria for hEDS or Hypermobile Spectrum Disorder (HSD) will receive aVNS (acoustic vagal nerve stimulation) therapy via filtered vocal music sound therapy using the Safe and Sound protocol (randomized 1:1 to active vs sham music; double blind study design)
  Interventions: Other: Acoustic vagal nerve stimulation (aVNS) treatment
- Treatment Arm B (ANS Dysfunction) (Experimental): (n=30) patients with concerns for ANS dysfunction (with or without hEDS) will receive auricular percutaneous vagal nerve stimulation (pVNS) therapy. Additional sub-study option: 15-20 subjects will undergo gastric MRI and (those who consent to it) will also participate in a biobank blood sample collection study.
  Interventions: Device: Percutaneous vagal nerve stimulation (pVNS) device

INTERVENTIONS:
Device: Percutaneous vagal nerve stimulation (pVNS) device — Subjects in Treatment Arm B will enter a six-week, prospective open label treatment trial with the FDA-approved and commercially available device IB-Stim. This is an ambulatory, neurostimulation device which consists of a battery powered, externally affixed generator with 4 wire leads attached to electrode/needle arrays affixed to the outer ear. The device delivers low voltage (3.2V) stimulation in alternating frequencies for a total of 5 days (around the clock).
  Other Names: percutaneous electrical nerve field stimulation
  Arms: Treatment Arm B (ANS Dysfunction)
Other: Acoustic vagal nerve stimulation (aVNS) treatment — All subjects receiving acoustic therapy via active VNS (aVNS; n=30) or sham VNS (sVNS; n=30) will enter a four-week, randomized, double-blind clinical trial during which they will listen to either computer altered/filtered vocal music (active treatment) that has been designed to stimulate vagal calming vs. regular non-filtered music (sham treatment). The stimuli will mirror the acoustic intervention known as the Safe and Sound Protocol. This protocol has been found to reduce auditory hypersensitivities and calming the autonomic nervous system by increasing vagal regulation of the heart via brainstem ventral vagal complex. The acoustic intervention may be played by an electronic device (i.e. smartphone, tablet, laptop, mp3) and delivered virtually with the help of trained coaches.
  Other Names: Safe and Sound Protocol
  Arms: Treatment Arm A (hEDS)

SUMMARY:
Hypermobile Ehlers-Danlos Syndrome (hEDS) is a connective tissue disorder characterized by hyperextensible skin, joint hypermobility and additional connective tissue manifestations. For unclear reasons, hEDS is associated with many gastrointestinal (GI) and autonomic nervous system (ANS) complaints such as postural orthostatic tachycardia syndrome (POTS). This study will address the clinical relationship between hEDS/Hypermobile Spectrum Disorders and autonomic regulation and see if there is a benefit of two forms of non-invasive vagal nerve stimulation therapies to reduce GI symptoms in hEDS and POTS. The study will also investigate plausible effects of these nerve stimulation therapies on gastric function and autonomic signaling.

DETAILED DESCRIPTION:
Hypermobile Ehlers-Danlos Syndrome (hEDS) is a connective tissue disorder characterized by hyperextensible skin, joint hypermobility and additional connective tissue manifestations. For unclear reasons, hEDS and Hypermobile Spectrum Disorders are associated with many gastrointestinal (GI) and autonomic nervous system (ANS) complaints such as postural orthostatic tachycardia syndrome (POTS). Symptoms are often disabling and associated with poor quality of life and high health care costs. The proposed research will address the following understudied areas: 1) the clinical relationship between hEDS and autonomic regulation, 2) the potential benefit of two forms of non-invasive vagal nerve stimulation (VNS) therapies in reducing functional GI symptoms in hEDS and POTS, and 3) plausible effects of these VNS therapies on gastric motor function and neurohormonal signaling.

Clinical reports document a high co-morbidity between autonomic disorders and hEDS. This prospective study will focus on three major clinical questions: 1) Are there reliable neurophysiological markers associated with hEDS that can provide insights into the 'neural mechanisms' resulting in multisystem co-morbidities? 2) Will innovative intervention techniques designed to enhance autonomic regulation via two non-invasive vagal nerve stimulation techniques (e.g., auricular and acoustic VNS) provide substantial symptom reduction and improve the hEDS patients' quality of life? 3) Can a novel gastric MRI technique capture gastric motor function abnormalities in adolescents with hEDS?

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-18 years old
* Children with functional upper GI complaints and clinical suspicion for hEDS or HSD as well as a Beighton score of at least 4/9
* Children with functional upper GI complaints and clinical suspicion for ANS dysfunction
* De-identified data from our prior studies (IRB #689519 and IRB #1064187) of patients with functional GI disorders who do NOT meet criteria for hEDS will be used as a comparison group
* Children who are English-speaking and lack other explanation for symptoms
* Children willing to participate and consent to this study (for children, have a parent willing to participate)

Exclusion Criteria:

A) Exclusion Criteria applying to all participants:

* Medically complex children or those who take a medication or suffer from a disease that can explain symptoms will be excluded from participation in the study.
* Adult subjects, children or their parents who have significant developmental delay (will be excluded due to difficulties in accurately completing the questionnaires and assessing symptoms)
* Patients with findings of organic disease such as peptic ulcer disease, H.pylori gastritis, celiac disease, inflammatory bowel disease, allergic disorders, metabolic disorder or any other chronic condition or medication that may cause chronic GI symptoms will be excluded from the study.
* Patients who are treated with a new drug affecting the central nervous system in the two weeks prior to enrollment will also be excluded.
* Pregnancy (evaluating MD screens patients as they normally would during a clinic visit (by questioning) and would only perform urine pregnancy test if clinically indicated (absence of menstrual period or other symptoms concerning for pregnancy)
* Chronic alcohol/illicit drug use and/or smoking.

B) Exclusion Criteria for subjects undergoing pVNS therapy:

* Severe dermatological condition or active infection of external or middle ear
* Implanted electrical device

C) Exclusion Criteria for subjects undergoing aVNS therapy:

* Hearing impaired
* Sight impaired without correction
* Seizure disorder

D) Exclusion Criteria for subjects undergoing gastric motor function sub-study:

* Patients with pacemakers, metal clips used in previous surgery or other device which are not compatible with MRI scanning
* Claustrophobia or inability to lie still in the scanner
* Orthodontic braces or permanent retainers
* Patients who are unable to tolerate noise produced by the MRI
* Egg allergy or anticipated inability to complete a standardized egg meal

E) Exclusion Criteria for subjects undergoing HepGI Biobank specimen collection sub-study:

* Bleeding disorder for the specific biopsies
* Recent antibiotic usage for fecal sample
* Significant anemia or clinical status which will not allow safe blood draw required for blood collection
* Refusal of blood collection or to provide DNA sample
* Inability or unwillingness on the individual (or parent/legal guardian) to provide clinical or family history.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gastrointestinal symptoms as assessed by the instrument Patient Assessment of upper Gastrointestinal Symptom Severity Index (PAGI-SYM) | Change from baseline total PAGI-SYM score at end of therapy (6 weeks)
  Instrument assessing upper gastrointestinal symptoms including symptoms of gastroparesis; score range 0-100 with higher scores indicating worse symptoms

SECONDARY OUTCOMES:
Change in gastric motor function as assessed by gastric MRI | Change from baseline at end of therapy (6 weeks)
  Dynamic gastric MRI measure of gastric accomodation as measured by gastric volume change in response to test meal. A greater gastric volume change indicates improved gastric accomodation.
Change in Body Perception Questionnaire (BPQ) total score | Change from baseline at end of therapy (6 weeks)
  Instrument assessing symptoms of autonomic reactivity; raw score range 0-130 with higher score indicating greater autonomic reactivity
Change in vagal efficiency measurements | Change from baseline at end of therapy (6 weeks)
  Metrics of vagal tone extracted from ECG R-R interval data measurements during postural challenges

CONTACTS AND LOCATIONS:
Overall Officials: Katja Kovacic, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castori M, Tinkle B, Levy H, Grahame R, Malfait F, Hakim A. A framework for the classification of joint hypermobility and related conditions. Am J Med Genet C Semin Med Genet. 2017 Mar;175(1):148-157. doi: 10.1002/ajmg.c.31539. Epub 2017 Feb 1. PMID 28145606
- [Background] Kovacic K, Chelimsky TC, Sood MR, Simpson P, Nugent M, Chelimsky G. Joint hypermobility: a common association with complex functional gastrointestinal disorders. J Pediatr. 2014 Nov;165(5):973-8. doi: 10.1016/j.jpeds.2014.07.021. Epub 2014 Aug 20. PMID 25151198
- [Background] Gazit Y, Nahir AM, Grahame R, Jacob G. Dysautonomia in the joint hypermobility syndrome. Am J Med. 2003 Jul;115(1):33-40. doi: 10.1016/s0002-9343(03)00235-3. PMID 12867232
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Porges SW, Davila MI, Lewis GF, Kolacz J, Okonmah-Obazee S, Hane AA, Kwon KY, Ludwig RJ, Myers MM, Welch MG. Autonomic regulation of preterm infants is enhanced by Family Nurture Intervention. Dev Psychobiol. 2019 Sep;61(6):942-952. doi: 10.1002/dev.21841. Epub 2019 Mar 13. PMID 30868570